CLINICAL TRIAL: NCT01082289
Title: A Phase 1, Open-Label, Drug-Drug Interaction Study to Determine the Effect of Repeated Dose Lurasidone 120 mg Administration on the Pharmacokinetics of Orally Administered Digoxin 0.25 mg in Patients With Schizophrenia or Schizoaffective Disorder.
Brief Title: Digoxin Drug-Drug Interaction With Lurasidone HCl
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group
Other Study IDs: D1050279
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2011-09

CONDITIONS: Schizophrenia
Keywords: Lurasidone; Schizophrenia; Latuda
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride

INTERVENTIONS:
Drug: Lurasidone

SUMMARY:
The objective of this study is to evaluate the pharmacokinetic profile of digoxin when administered alone and when administered with repeated dose of lurasidone 120mg.

ELIGIBILITY:
Inclusion Criteria:

* Male and female 18 to 65 years of age
* BMI >= 19.5 and <= 37 kg/m2
* No clinically relevant abnormal laboratory values

Exclusion Criteria:

* History or presence of renal or hepatic insufficiency
* Participated in a clinical trial in the past 30 days
* Use of con meds that prolong the QT/QTc taken within 28 days prior to study drug administration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marina Bussel, MD, Principal Investigator — California Clinical Trials
Locations (1):
- California Clinical Trials, Culver City, California, United States